CLINICAL TRIAL: NCT02747446
Title: Effects of a Dietary Honey or Isomolar Fructose:Glucose Mixture on Glucose Tolerance and Blood Lipid Profile in Healthy Male Volunteers
Brief Title: Metabolic Effects of Honey or Fructose:Glucose Mixtures
Acronym: HONEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luc Tappy, MD (Other)
Collaborators: Agroscope Liebfeld Posieux, Liebfeld-Bern Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 154/12
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: fructose, triglyceride, oral glucose tolerance
MeSH Terms: interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Honey (Experimental): added sugar: diet with 25% acacia honey
  Interventions: Dietary Supplement: added sugar
- Fructose:glucose mixture (Experimental): added sugar: Diet with 25% energy as a fructose:glucose mixture
  Interventions: Dietary Supplement: added sugar
- control (No Intervention): no intervention: Diet with 45% starch and no honey or added sugars

INTERVENTIONS:
Dietary Supplement: added sugar — isocaloric substitution of added sugars (honey or FG) for starch
  Arms: Fructose:glucose mixture; Honey

SUMMARY:
The metabolic effects of 7-day weight-maintenance diets containing 10% total energy as acacia honey or a fructose:glucose mixture will be assessed in a group of healthy male volunteers. Primary outcome is plasma total triglyceride concentrations after ingestion of standardized breakfast and lunch containing 25% energy as honey or fructose:glucose mixture; secondary outcome is glucose tolerance and suppression of endogenous glucose production after ingestion of 75 g glucose. Results obtained with 10% honey and 10% fructose: glucose mixture diets will be compared to results obtained with a weight-maintenance, isocaloric diet in which starch is substituted for honey or fructose:glucose mixture

DETAILED DESCRIPTION:
Eight health males volunteers will be studied three times in a randomized order

* Honey: volunteers will be fed a weight-maintenance diet containg 5% sugars, 20% starch, 25% acacia honey, 35% fat and 15% protein during 6 days (day 1-6); On day 7, their plasma metabolites and hormones concentrations will be monitored over 10 hours during which they will receive a breakfast and a lunch containing honey; on day 8, they will have a 75g oral glucose4 + 375 mg 13C-labelled glucose tolerance test, and their plasma glucose and insulin concentrations will be monitored over 4 hours; glucose kinetics will be measured by 6,6 deuterated glucose
* FG: volunteers will be fed a weight-maintenance diet containg 5% sugars, 20% starch, and 25% of a fructose:glucose mixture matching the composition of acacia honey, 35% fat and 15% protein during 6 days (day 1-6); On day 7, their plasma metabolites and hormones concentrations will be monitored over 10 hours during which they will receive a breakfast and a lunch containing fructose and glucose; on day 8, they will have a 75g oral glucose + 375 mg 13C-labelled glucose tolerance test, and their plasma glucose and insulin concentrations will be monitored over 4 hours; glucose kinetics will be measured by 6,6 deuterated glucose
* Control: volunteers will be fed a weight-maintenance diet containg 5% sugars, 45% starch, 35% fat and 15% protein during 6 days (day 1-6); On day 7, their plasma metabolites and hormones concentrations will be monitored over 10 hours during which they will receive a breakfast and a lunch with no added sugar; on day 8, they will have a 75g oral glucose + 375 mg 13C-labelled glucose tolerance test, and their plasma glucose and insulin concentrations will be monitored over 4 hours; glucose kinetics will be measured by 6,6 deuterated glucose

ELIGIBILITY:
Inclusion Criteria:

* health volunteer

Exclusion Criteria:

* BMI < 19.5
* BMI > 25
* Smoker
* Any disease
* current treatment with any drug

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
plasma total triglyceride profile | 7-day dietary intervention
  plasma triglyceride concentrations measured before and after ingestion of a breakfast and a lunch

SECONDARY OUTCOMES:
glucose tolerance | 7-day dietary intervention
  plasma glucose and insulin concentration and suppression of endogenous glucose production after ingestion of 75 g glucose

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- CHUV-clinical research center, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided